CLINICAL TRIAL: NCT02892279
Title: Sympathetic Nerve Activation Evoked by Diesel Exhaust Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Jenny Bosson, MD, PhD, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Umu-2016-57-31
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Microneurography; Air pollution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diesel exhaust exposure (Experimental): A single arm study in which first a baseline muscle sympathetic nerve activity (MSNA) is recorded with and without an exposure mask. When measurements have been secured exposure to dilute diesel exhaust will start.
  Interventions: Other: Diesel exhaust exposure

INTERVENTIONS:
Other: Diesel exhaust exposure — Evaluation of sympathetic nervous system activity as assessed by microneurography recording during an acute exposure to dilute diesel exhaust via mask.

SUMMARY:
The adverse effects of air pollution on cardiovascular and respiratory health have been demonstrated in an extensive series of epidemiological, observational and experimental studies. In the current project the investigators aim to determine whether an acute exposure to diesel exhaust causes impacts on sympathetic nervous system activation in healthy volunteers.

DETAILED DESCRIPTION:
Brief as well as chronic exposures to air pollution have been linked with increases in cardiovascular morbidity and mortality. Evidence suggests that the strongest associations between air pollution exposure and adverse cardiovascular effects are found for combustion-derived particulate matter, especially in the fine and ultrafine ranges such as is found in diesel engine emissions. Despite a greater understanding of the cardiovascular effects of air pollution, the underlying mechanism through which exposure to fine particulate air pollution alters vascular function has yet to be determined. Microneurography is a method that records nerve impulse traffic in human peripheral nerves, allowing for the assessment of sympathetic nervous activity. The current study will employed microneurography techniques to evaluate autonomic function in association with inhaled air pollution exposure in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (normal ECG, lung function, blood sample, clinical examination)

Exclusion Criteria:

* Metabolic disease
* Cardiovascular disease
* Respiratory disease
* BMI ≥ 30
* Use of psychoactive medication
* Infection within 2 weeks of the study
* Smokers or regular snus usage

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Microneurography | 1 hour
  Microneurography recording of muscle sympathetic nervous system activity

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Bosson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Dept of Medicine, Lung and Allergy section, University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rankin GD, Kabele M, Brown R, Macefield VG, Sandstrom T, Bosson JA. Acute Exposure to Diesel Exhaust Increases Muscle Sympathetic Nerve Activity in Humans. J Am Heart Assoc. 2021 May 18;10(10):e018448. doi: 10.1161/JAHA.120.018448. Epub 2021 May 4. PMID 33942621